CLINICAL TRIAL: NCT05643157
Title: Structure and Function of Retinal Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kristen Bowles Johnson, Post Doctoral Researcher, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18287
Record Dates: First submitted 2022-11-08; First posted 2022-12-08 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-06

CONDITIONS: Retinal Toxicity
Keywords: retinal toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Retinal Disease (Experimental): Subjects with either retinal toxicity or inherited retinal degeneration will undergo multimodal clinical imaging and Adaptive Optics Optical Coherence Tomography (AO-OCT) imaging at each study visit to document regions of disease and healthy retina over time.
  Interventions: Device: Adaptive Optics - Optical Coherence Tomography (AO-OCT) retinal imaging

INTERVENTIONS:
Device: Adaptive Optics - Optical Coherence Tomography (AO-OCT) retinal imaging — AO-OCT used in this study is an investigational OCT imaging system. . In this instrument, ocular aberration sensing and correction is achieved with a Shack-Hartmann wavefront sensor (SHWS) and deformable mirror, respectively. A pupil camera and fixation target are used to position the participant's head and eye for scanning a particular retinal region within 15 degrees of the fovea. Data collected generally includes AO-OCT volume videos and SHWS measurements of ocular aberrations.

SUMMARY:
Current clinical cameras do not allow clinicians to see the cells of the retina. This study will evaluate a new electronic camera's ability to image the human retina in finer detail.

DETAILED DESCRIPTION:
This research study will (1) test the ability of a new electronic camera developed in Dr. Miller's laboratory to collect extremely sharp volumetric images of the retina in human subjects, and (2) use the camera for addressing fundamental questions about how disease progresses in the eye. This new camera integrates cutting-edge technologies in adaptive optics (AO) and optical coherence tomography (OCT) that enable the camera to capture sharp images. However, many aspects of the camera are already employed in clinical instruments used routinely by eyecare practitioners worldwide. The objective of our study is to find out (1) whether the AO-OCT camera will allow researchers to observe and quantify finer detail in the retina than current clinical cameras, and (2) whether this finer detail is useful for understanding the progression of disease in the eye.

To address the second objective, the study will look at two subgroups of retinal disease. The first is age-related macular degeneration (AMD), a leading cause of blindness in the developed world. Because this disease is difficult to study directly as it takes years to progress, we will study it indirectly using subjects with a form of retinal toxicity that exhibits a retinal phenotype similar to that of AMD but progresses on a much faster time scale. The second disease subgroup is inherited retinal degeneration that affects as many as 1 in every 2,000 people worldwide. For this subgroup, the researchers will test the exquisite sensitivity of the AO-OCT imaging system to detect minute changes in disease progression over short periods of time covering weeks and months.

ELIGIBILITY:
Inclusion Criteria:

* Retinal disease of either inherited retinal degeneration or retinal toxicity

Exclusion Criteria:

* Ocular media opacities
* High refractive error
* Pupil dilation imposes a risk to ocular health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of photoreceptor and retinal pigment epithelium (RPE) cell layers | 2 years
  Images of the photoreceptor and RPE cell layers taken with clinical instruments and the AO-OCT will be compared.
RPE cell morphology changes | 2 years
  Images will be used to determine the changes in RPE cell morphology in regions of healthy and diseased retina (in subjects with retinal disease).
Cone Photoreceptor Dysfunction | 2 years
  Images will be used to determine changes in cone photoreceptor dysfunction and death

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Optometry, Bloomington, Indiana, United States